CLINICAL TRIAL: NCT01074801
Title: An Open-label, Randomised, 2-period Cross-over Study to Assess the Efficacy and Safety of 36-hour Closed-loop Glucose Control in Comparison With Conventional Subcutaneous Insulin Pump Treatment in Adolescents With Type 1 Diabetes
Brief Title: Closing the Loop for 36 Hours in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Stephen Kelleher, Cambridge University Hospitals NHS Foundation Trust and University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DAN01
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2011-04-06 (Estimated); Status verified 2010-02

CONDITIONS: Type 1 Diabetes
Keywords: Closed-loop systems; day-and-night glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed-loop (Active Comparator): Subcutaneous insulin delivery to be adjusted according to the computer-based algorithm advice, based on subcutaneous glucose readings
  Interventions: Other: Closed-loop insulin delivery
- Control arm (Active Comparator): Subcutaneous insulin delivery to be administered according the standard insulin pump settings
  Interventions: Other: Standard insulin pump treatment

INTERVENTIONS:
Other: Closed-loop insulin delivery — Basal subcutaneous insulin delivery to be adjusted at 15min cycles according to the computer-based algorithm advice.
  Arms: Closed-loop
Other: Standard insulin pump treatment — Subcutaneous insulin delivery to be performed based on subjects' standard treatment
  Arms: Control arm

SUMMARY:
High variability of blood sugar levels and high incidence of night-time hypoglycaemia (low blood sugar) in young people with type 1 diabetes (T1D) make achieving the treatment goals in this population extremely challenging.

Our ongoing research focuses on the development of a closed-loop glucose control in children and adolescents with T1D. The three components of the closed-loop system are a continuous glucose monitor, an insulin pump, and a computer-based algorithm. The studies performed thus far evaluated the efficacy and safety of overnight closed-loop glucose control. The results showed that overnight closed-loop improved control of blood glucose and prevented nocturnal hypoglycaemia, as compared to the conventional insulin pump therapy. The next objective is to evaluate the efficacy and safety of closed-loop insulin delivery over a prolonged time period, including the daytime, when normal living activities occur. This will pave the way for a more comprehensive use of closed loop systems to control glucose levels in T1D.

The present study adopts an open-label, randomised, 2-period cross-over design whereby the safety and efficacy of closed-loop insulin therapy will be compared with the conventional insulin pump therapy in 12 adolescents with T1D. Participants aged 12 to 18 years will be randomised for two 36 hour studies in a clinical research facility, during which glucose levels will be controlled by either the computer-based closed-loop algorithm (intervention arm) or by conventional insulin pump therapy (control arm). During both studies participants will perform normal daily activities, i.e. playing, reading, snacking and physical activity. On both occasions, the Actiheart, a combined heart rate and movement sensor will be used to accurately quantify each subject's individual physical activity energy expenditure during the 36 hour study period and for 36 hours of free living during weekday.

DETAILED DESCRIPTION:
The study is an open-label, randomised, 2-period crossover study comparing the closed-loop insulin therapy with the conventional insulin pump therapy in 12 adolescents with type 1 diabetes.

Subjects who consented to take part in the study will attend the Clinical Research Facility on two occasions, each lasting 36 hours. Approximately 1-3 days prior to each Study Visit, a subcutaneous continuous glucose monitoring (CGM) device will be inserted.

On each Study Visit subjects will arrive between 17:30 and 18:00 and will stay in the clinical research facility for two nights.

Shortly after arrival the subjects will have Actiheart monitor fitted and a cannula inserted into a vein of one arm for blood sampling purposes. Blood sampling for plasma glucose and plasma insulin will start at 18:30 and will be carried out at 30 minutes intervals during the day and at 60min intervals during the night throughout the study period. Plasma glucose measurements will be done in real time every 30min during the day and every 60min during the night except when when plasma glucose < 3.5mmol/L or following treatment for hypoglycaemia, when the measurements will be carried out every 15 minutes.

On Study Visit 1 the subjects will be randomised on arrival to receive either the conventional insulin pump therapy or the closed-loop intervention. At 18:30 subjects will perform 5 to 10 minutes exercise on a bicycle to determine the settings needed to achieve a heart rate of 140 bpm corresponding to an exercise level at 55%60% of peak VO2. In the closed-loop intervention arm the insulin pump therapy will be driven by the computer-based algorithm from 19:30 until the end of the study. The basal insulin infusion rate on the insulin pump will be adjusted manually at 15min intervals following the computer-based algorithm advice. During the control arm, the subject will carry on with their usual insulin pump regimen. In both groups CGM will be continued throughout the whole of the study period. Subjects who completed Study Visit 1 will cross over to the alternative Study Visit schedule after an interval of 1 to 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The subject is between 12 and 18 years of age (inclusive)
* The subject has had type 1 diabetes, as defined by WHO for at least 1 year or is confirmed C-peptide negative
* The subject will have been on insulin pump for at least 3 months, with good knowledge of insulin self-adjustment
* HbA1c ≤ 12% based on analysis from central laboratory

Exclusion Criteria:

* Non-type 1 diabetes mellitus including those secondary to chronic disease
* Any other physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results
* Current treatment with drugs known to interfere with glucose metabolism such as systemic corticosteroids, non-selective beta-blockers and MAO inhibitors
* Known or suspected allergy against insulin
* Subjects with clinical significant nephropathy, neuropathy or proliferative retinopathy as judged by the clinician
* Total daily insulin dose >= 2 IU/kg
* Postmenarchal girls who are pregnant or intending to become pregnant or are breastfeeding
* Any coexisting cardiac and respiratory condition (including asthma)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is time spent with plasma glucose concentration in the target range (3.9-10.0 mmol/L) between 24:00 on Day 1 to 08:00 on Day 3. | 32 hours

SECONDARY OUTCOMES:
Secondary outcomes will include: (i) Total and basal insulin delivery between 24:00 on Day 1 and 08:00 on Day 3 (36 hours) (ii) CGM glucose levels between 24:00 on Day 1 and 08:00 on Day 3 (36 hours) | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Wellcome Trust Clinical Research Facility, Addenbrooke's Hospital, Cambridge, United Kingdom